CLINICAL TRIAL: NCT00726063
Title: A Prospective Randomized-controlled Evaluation of Nanotite and Osseotite Surfaced Implant Performance in Graduate Student Programs
Brief Title: A Prospective Study Evaluating the Performance of Nanotite Osseotite Implants When Placed by Graduate Student Programs
Acronym: CollegeBowl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2613
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Tooth Disease; Partial Edentulism
Keywords: dental implants; Nanotite implant; Osseotite implants; multicenter; randomized; clinical study; partial edentulism; prosthesis
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Intervention Model Description: implant types were randomized- 2 different surface treatments
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nanotite implant (Experimental): Nanotite dental implant
  Interventions: Device: Nanotite dental implant
- Osseotite implant (Active Comparator): Osseotite dental implant
  Interventions: Device: Osseotite dental implant

INTERVENTIONS:
Device: Nanotite dental implant — Nanotite root form titanium dental implant
  Other Names: Nanotite endosseous dental implant
  Arms: Nanotite implant
Device: Osseotite dental implant — Osseotite Root form titanium dental implant
  Other Names: Osseotite endosseous dental implant
  Arms: Osseotite implant

SUMMARY:
This study will evaluate the contributions of the Nanotite implant design when used by graduate students in their first year of placing implants.

DETAILED DESCRIPTION:
This multicenter, prospective, randomized-controlled study will compare the performance of the Nanotite vs. the standard Ossotite implants when placed by graduate students with little or no prior experience. Enrolled patients will have the study site(s) randomized to either a Nanotite (test) or an Osseotite (control) implant. The manner of treatment observed at the participating center will be followed for this study.

Study Hypothesis: The performance of the Nanotite implant in this study will be no different than or superior to that of the Osseotite implant placed during the early period of graduate student training.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and of any race, 18 years of age or older
* patients for whom a decision has already been made to use dental implants for treating edentulism in the mandible or maxilla

Exclusion Criteria:

* patients who are known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Reddy, DMD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 165 patients are expected to be enrolled across all centers, with enrollment efforts beginning in August 2008. Enrollment period remained opent until December 2010.
Pre-assignment Details: Pre-treatment included a screening visit (enroll those meeting all protocol inclusion criteria), signing informed consent, and pre-surgical data collection. Patients returned for implant placement surgery, followed by restorative activities.
Groups:
- Nanotite Implant: Nanotite dental implant
  Nanotite dental implant : Nanotite root form titanium dental implant
- Osseotite Implant: Osseotite dental implant
  Osseotite dental implant : Osseotite Root form titanium dental implant
Period: Overall Study
Arm/Group | Nanotite Implant | Osseotite Implant
Started | 122 (Number of implants= 239) | 119 (Number of implants= 246)
Completed | 113 (Number of implants =230) | 112 (Number of implants = 239)
Not Completed | 9 | 7
Not completed — Adverse Event | 9 | 7

BASELINE CHARACTERISTICS:
Population: Nanotite implants = 239 Osseotite implants = 246
Groups:
- Total: Total of all reporting groups
Arm/Group | Nanotite Implant | Osseotite Implant | Total
Number analyzed (Participants) | 122 | 119 | 241
Age, Categorical [Count of Participants; unit: Participants] — Overall number of Nanotite implants = 239 Overall number of Osseotite implants = 246 Nanotite implants in <18 yrs = 1 Nanotite implants in 18-65 = 163 Nanotite implants in >65 = 75 Osseotite implants in <18 yrs = 0 Osseotite implants in 18-65 = 173 Osseotite implants in >65 = 73
  Participants
    <=18 years | 1 | 0 | 1
    Between 18 and 65 years | 61 | 63 | 124
    >=65 years | 60 | 56 | 116
Sex: Female, Male [Count of Participants; unit: Participants] — Overall number baseline implants Nanotite= 239 Overall number baseline implants Osseotite = 246 Nanotite implants in Females = 116 Nanotite implants in Males = 123 Osseotite implants in Females = 120 Osseotite implants in Males = 126
  Participants
    Female | 61 | 64 | 125
    Male | 61 | 55 | 116

OUTCOME MEASURES:

1. Primary Outcome: Integration Success of the Implant
Time Frame: 1 year
Population: Number of implants surviving (lack of mobility) at the end of the study (time of analysis)
Measure: Number; unit: implants
Units Other Than Participants: Implants
Arm/Group | Nanotite Implant | Osseotite Implant
Number analyzed (Participants) | 122 | 119
Number analyzed (Implants) | 239 | 246
implants | 230 | 239

ADVERSE EVENTS:
Time Frame: Adverse events are collected and reported throughout the duration of the study, an average of 2 years.
Description: Adverse event data is collected by patient questioning,visual examination, and radiologic assessment of patient's treatment area each study event visit.
Arm/Group | Nanotite Implant | Osseotite Implant
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/119
Other Adverse Events (participants affected / at risk) | 9/122 | 7/119
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nanotite Implant (N=122) | Osseotite Implant (N=119)
Loss of integration of implant (Surgical and medical procedures) | 9 (9) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall furnish SPONSOR with a copy of any proposed publication thirty (30) days prior to submission for publication for review and comment. SPONSOR may request PI to delay publishing such proposed publication for a maximum of an additional sixty (60) days in order to protect the potential patentability of any invention described therein.